CLINICAL TRIAL: NCT05233709
Title: The Effect of Ovotransferrin and Lactoferrin on Iron Absorption From Ferrous Sulfate in Adult Women With Non-anemic Iron Deficiency: Stable Isotope Study
Brief Title: The Effect of Ovotransferrin and Lactoferrin on Iron Absorption From Ferrous Sulfate in Adult Women
Acronym: OTf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OTf
Record Dates: First submitted 2021-10-29; First posted 2022-02-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OTf + FeSO4 (Other): OTf + FeSO4 - This is the experimental arm where Ferrous sulfate will be given to the participants along with apo-Ovotransferrin, a potential iron absorption enhancer. They will be given as solutions that will be spread on bread with butter and honey, a breakfast meal.
  Interventions: Dietary Supplement: FeSO4 + OTf
- Lf+ FeSO4 (Other): Lf + FeSO4 - This is the experimental arm where Ferrous sulfate will be given to the participants along with lactoferrin, a potential iron absorption enhancer. They will be given as solutions that will be spread on bread with butter and honey, a breakfast meal.
  Interventions: Dietary Supplement: FeSO4 + Lf
- FeSO4 (Other): FeSO4 - This is the control arm where Ferrous sulfate will be given in the form of a solution that will be spread on bread with butter and honey, as a breakfast meal
  Interventions: Dietary Supplement: FeSO4

INTERVENTIONS:
Dietary Supplement: FeSO4 + OTf — OTf (apo ovotransferrin) + FeSO4
  Arms: OTf + FeSO4
Dietary Supplement: FeSO4 + Lf — Lf (lactoferrin) + FeSO4
  Arms: Lf+ FeSO4
Dietary Supplement: FeSO4 — Ferrous sulfate
  Arms: FeSO4

SUMMARY:
OTf is a monomeric glycoprotein of 686 amino acid residues and, as a member of the transferrin family, folds into two homologous globular lobes, each containing a single reversible Fe3 + binding site located within the interdomain cleft of each lobe. A comparison of apo (metal-free) and holostructures shows that iron binding or release in OTf occurs via a mechanism that involves opening or closing domains. human lactoferrin, transferrin, and OTf share the same reversible iron binding mechanism. Lactoferrin (Lf) is a 77 kDa glycosylated protein highly concentrated in human and bovine milk and can exist in an apo (metal free) state or can bind two ferric ions with very high affinity (k = 1022 M-1) forming holo-Lf . It has been recently reported that the addition of apo-Lf to a test meal containing FeSO4 significantly increased (+56%) iron absorption in young infants [19]. Despite these positive results in infants, to our knowledge, the ability of Lf to improve iron absorption from FeSO4 has not yet been assessed in adult women.

OTf and Lf will be tested as iron absorption enhancers by comparing the fractional iron absorption with that of FeSO4, the most widely used iron supplement. This study will provide information on how to improve iron absorption.In a randomized single-blind crossover study, the iron bioavailability is determined by means of stable iron isotope technology via the incorporation of stable isotopes from intrinsically labeled compounds into the erythrocytes 14 days after the study product.

DETAILED DESCRIPTION:
Iron deficiency remains a major public health problem in both developed and developing countries. At present, iron deficiency is mostly combated with iron supplements in the form of iron salts, especially iron sulfate. Iron salts are absorbed via the nonhemic iron route via the DMT-1 receptor, the rate of absorption being 20% of the total iron content. The dietary supplement industry tries to counteract this problem and to supply the required amount of iron by increasing the iron concentration in the dietary supplements in order to compensate for the low absorption rate. However, the high dosage of iron leads to side effects. It would be more effective to maximize iron absorption rather than a high dose of iron. Chicken protein ovotransferrin (OTf) is recognized as an iron-binding protein and a member of the transferrin family. OTf has amino acid sequences that are identical to chicken serum transferrin and shows approximately 50% homology with mammalian transferrin and lactoferrin. Despite its iron binding properties and safety for human consumption, no studies have evaluated OTf as an enhancer of iron absorption in humans.

OTf is a monomeric glycoprotein of 686 amino acid residues and, as a member of the transferrin family, folds into two homologous globular lobes, each containing a single reversible Fe3 + binding site located within the interdomain cleft of each lobe. A comparison of apo (metal-free) and holostructures shows that iron binding or release in OTf occurs via a mechanism that involves opening or closing domains. human lactoferrin, transferrin, and OTf share the same reversible iron binding mechanism.

Lactoferrin (Lf) is a 77 kDa glycosylated protein highly concentrated in human and bovine milk and can exist in an apo (metal free) state or can bind two ferric ions with very high affinity (k = 1022 M-1) forming holo-Lf . There are various studies that show the iron bioavailability of intrinsically labeled holo-Lf and apo- Lf and FeSO4. Lf appears to be a good source of bioavailable iron in both infants and in adults. Whether this is due to iron absorption through the Lf receptor and/or due to iron released from Lf joining the common non-heme iron pool and being subsequently absorbed, remains uncertain. The high affinity of OTf for iron (∼1030 M-1) at pH 7.5 implies that in presence of apo-OTf, iron will be sequestered. Lf also possesses the ability to bind iron (binding constants of ∼1022-1024 M-1) and retain it at lower pH. This difference in iron binding capacity, however, is not sufficient to establish conclusive statements regarding the activity of OTf in iron absorption.

It has been recently reported that the addition of apo-Lf to a test meal containing FeSO4 significantly increased (+56%) iron absorption in young infants. Despite these positive results in infants, to our knowledge, the ability of Lf to improve iron absorption from FeSO4 has not yet been assessed in adult women. Furthermore, despite its iron-binding properties and safety for human consumption, to the best of our knowledge, no studies have assessed OTf as an enhancer of iron absorption in humans. Therefore the use of OTf and Lf as iron absorption enhancers by comparing fractional iron absorption with that of FeSO4, the most commonly used iron supplement is investigated. This study will provide information regarding iron absorption enhancement, as well the behavior of OTf and Lf in adult women.

OTf and Lf will be tested as iron absorption enhancers by comparing the fractional iron absorption with that of FeSO4, the most widely used iron supplement. This study will provide information on how to improve iron absorption.In a randomized single-blind crossover study, the iron bioavailability is determined by means of stable iron isotope technology via the incorporation of stable isotopes from intrinsically labeled compounds into the erythrocytes 14 days after the study product.

Participants are given OTf, Lf and iron sulfate solutions. To quantify this, stable iron isotopes are used as marker substances. Stable isotopes exist in nature and in our body and there are no risks associated with their ingestion. No changes in the iron status of the subjects are expected during the study.35 women of childbearing age are being recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* female aged between 18-45 years old;
* SF <25 µg / L;
* BMI 18.5-24.9 kg / m2;
* weight <70 kg;
* signed informed consent;
* Able to communicate and comprehend English language.

Exclusion Criteria:

* Anemic (Hb <12 g / dL);
* inflammation (CRP> 5 mg / L);
* chronic digestive, renal and / or metabolic disease;
* chronic medications (except for oral contraceptives);
* use of vitamin, mineral and pre- and / or probiotic supplements in the previous 2 weeks and during the course of the study;
* blood transfusion, blood donation or significant blood loss over the past 4 months;
* difficulties with blood sampling;
* antibiotic treatment in the previous 4 weeks before the start of the study and during the course of the study;
* known hypersensitivity to egg;
* pregnancy (tested in serum at screening) or intention to become pregnant during the course of the study;
* lactation up to 6 weeks before study initiation;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption | Day 19th of the study
  The primary outcome is iron bioavailability (as measured by erythrocyte incorporation of the stable isotope labels) from the 2 different conditions in the standardized test meals.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | Screening (-14,) day 1 and day 19th
  Iron status marker
Serum ferritin (SF) | Screening (-14,) day 1 and day 19th
  Iron status marker
Serum transferrin receptor (sTfR), | Screening (-14,) day 1 and day 19th
  Iron status marker
C-reactive protein (CRP) | Screening (-14,) day 1 and day 19th
  Inflammation status

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Rigutto-Farebrother, PhD, Principal Investigator — Laboratory of Human Nutrition ETH Zürich
Locations (1):
- ETH Zurich, Laboratory of Human Nutrition, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No